CLINICAL TRIAL: NCT03958968
Title: Impact of Exposure to Cosmetics on Sensitive Skin
Acronym: SENSICOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SENSICOS (29BRC18.0078)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-01

CONDITIONS: Sensitive Skin; Cosmetic Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The concept of sensitive or reactive skin was evoked in 1947 and developed in the 1970s and is now widely recognized. The international pruritus society has proposed an international consensus definition: sensitive skin is defined as a syndrome manifested by the occurrence of unpleasant sensations (tingling, burning, pain, pruritus, tingling) in response to stimuli that normally do not not cause such sensations. The triggering factors can be cosmetics, water, cold, heat, temperature variations, wind ... etc.

The physiopathological mechanisms are debated and several hypotheses exist. Sensitive skin can be considered as a decrease of the threshold of cutaneous tolerance. Sensitive skin is linked to abnormalities of the cutaneous nervous system, which becomes hyper-reactive. This hyperreactivity can be modulated by multiple factors. Exposure to cosmetics could be one of the main triggers for sensitive skin, especially for women. This can be explained by the wide use of cosmetics (in France women apply an average of 16 different cosmetics per day), by overconsumption of cosmetics, by exposure to potentially irritating ingredients. Sensitive skin would be less tolerant to the frequent and prolonged use of cosmetics. However, no precise information is available on the actual consumption of cosmetic products in the population with sensitive skin, in particular no data exists concerning the type of products used, the criteria of choice of products, the daily number of products used. and the ingredients contained in these cosmetics

DETAILED DESCRIPTION:
Objectives are:

To compare the consumption of cosmetics qualitatively and quantitatively in a group of subjects with sensitive skin in the face and scalp, with a group of subjects with non-sensitive skin Study of triggers of sensitive skin Localization of sensitive skin in the face Resonance of sensitive skin Duration of onset of skin sensitivity after application of the cosmetic Use of organic products, formulated for sensitive skin, for children Shopping venues for cosmetics Advice from a professional for the purchase of cosmetics Impact of sensitive skin on the use of cosmetics Budget dedicated to the purchase of cosmetics

ELIGIBILITY:
Inclusion Criteria:

Women Between 18 and 65 years old -

Exclusion Criteria:

Men Less than 18 years old More than 65 years old Skin disease on the face: acne, rosacea, eczema Refusal to participate

-

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 150 persons
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Comparison of cosmetics use between subjects with and without sensitive skin | during the inclusion visit
  Ingredients contained in the cosmetics, type of products used and frequencies of use between a group of subjects with sensitive skin and a group without sensitive skin

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Laboratory Interaction Neurons Keratinocytes, Brest
  - Laboratory LINK, Brest